CLINICAL TRIAL: NCT01308294
Title: Vaccination of Melanoma Patients (Stage II-IV) With ImmuFact IMP321, Tumor Antigenic Peptides and Montanide
Brief Title: Immunotherapy of HLA-A2 Positive Stage II-IV Melanoma Patients
Acronym: LAG-3/IMP321
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low enrollment rate
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Immutep S.A.S. (Industry)
Responsible Party: Principal Investigator, Prof Olivier Michielin, M.D., Ph.D., Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P009-2010DR1082
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Results first posted 2020-03-20 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Melanoma
Keywords: Melanoma; Stage II-IV; Immunotherapy; Vaccination; HLA class I and II tumor-specific peptides; IMP321; Montanide ISA-51
MeSH Terms: conditions — Melanoma | interventions — soluble LAG-3 protein, human; Monatide (IMS 3015)

STUDY DESIGN:
Intervention Model Description: open label, non comparative study in patients suffering from stage II, III or IV melanoma
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 vaccine injections in 1 limb (Experimental): 9 patients initially planned: patients received peptides with IMP321/LAG-3Ig and Montanide in 2 injections sites at 5 cm distance from each other 2 vaccine injections in same limb (vaccine 1 : NY-ESO-1, MAGE-3.A2, NA-17 peptides + IMP321 + Montanide) (vaccine 2 : Melan-A, MAGE-A3-DP4 peptides + IMP321 + Montanide)
  Interventions: Biological: 2 vaccine injections in 1 limb
- 2 vaccine injections in distinct limbs (Experimental): Groupe2: 2 vaccine injections in different limb should include 9 patients that were initially planned: patients received the same vaccine in 2 syringes injected each in a distinct limb (vaccine 1: NY-ESO-1, MAGE-3.A2, NA-17 peptides + IMP321 + Montanide) (vaccine 2: Melan-A, MAGE-A3-DP4 peptides + IMP321 + Montanide)
  Interventions: Biological: 2 vaccine injections in distinct limbs
- 2 "vaccine injections" in distinct limbs (Experimental): Groupe3: 2 vaccine injections in distinct limb should include 9 patients that were initially planned; due to premature trial termination, no patients could be enrolled. Patients of this group should have received the same vaccine but without the MHC class II peptide (MAGE-A3)
  Interventions: Biological: 2 "vaccine injections" in distinct limbs

INTERVENTIONS:
Biological: 2 vaccine injections in 1 limb — Participants receive the vaccine separated in 2 syringes with syringe 1 containing NA-17, MAGE-3.A2 and NY-ESO-1 peptides with IMP321/LAG3 ± Montanide, and syringe 2 containing Melan-A and MAGE-A3-DP4 peptides with IMP321/LAG-3 ± Montanide. The content of each syringe is injected s.c. in the same limb at about 5 cm distance from each other.
  Other Names: vaccine1: NY-ESO-1,MAGE-3.A2, NA-17, IMP321, Montanide; vaccine 2: Melan-A, MAGE-A3-DP4 , IMP321, Montanide
  Arms: 2 vaccine injections in 1 limb
Biological: 2 vaccine injections in distinct limbs — Participants receive the vaccine separated in 2 syringes with syringe 1 containing NA-17, MAGE-3.A2 and NY-ESO-1 peptides with IMP321/LAG3 ± Montanide, and syringe 2 containing Melan-A and MAGE-A3-DP4 peptides with IMP321/LAG-3 ± Montanide.The content of each syringe is injected s.c. in different limbs.
  Other Names: vaccine 1: NY-ESO-1, MAGE-3.A2, NA-17,IMP321, Montanide; vaccine 2: Melan-A, MAGE-A3-DP4, IMP321, Montanide)
  Arms: 2 vaccine injections in distinct limbs
Biological: 2 "vaccine injections" in distinct limbs
  Other Names: vaccine 1: NY-ESO-1, NA-17, IMP321, Montanide; vaccine 2: Melan-A, NA-17, IMP321, Montanide
  Arms: 2 "vaccine injections" in distinct limbs

SUMMARY:
The purpose of this study is to determine whether vaccination with tumor antigenic peptides and both IMP321/LAG-3 and Montanide adjuvants can induce an immune response in melanoma patients and to assess the safety and tolerability of this vaccination. Tumor responses following this vaccination will also be documented.

DETAILED DESCRIPTION:
The primary objective of this study is:

* to evaluate melanoma antigen specific immune response induced by this vaccination with tumor antigenic peptides derived from MAGE-A3 (Melanoma Antigen family A3) (MHCI: MAGE-A3.A2 and MHCII: MAGE-A3.DP4), NY-ESO-1 (New York Esophageal squamous cell carcinoma antigen-1), Melan A (analog ELA and native EAA) and NA-17A with IMP321 (ImmuFact)/ LAG-3Ig (Lymphocyte activation gene-3 immunoglobulin-like domains) as adjuvant/immunostimulant, formulated with Montanide ISA-51.
* to assess the safety and tolerability of this vaccination

The secondary objective is to document tumor responses in patients following this vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage II, III or IV melanoma patients.
* Tumor expression of Melan-A.
* Human leukocyte antigen-A2 (HLA-A2) positive.
* Expected survival of at list 3 months.
* Karnofsky scale performance status of 70 % or more.
* Age ≥ 18 years.
* Able to give a written informed consent.
* The following laboratory results:

Hemoglobin ≥ 100g/L, Neutrophil count ≥ 1.5 x 109/L, Lymphocyte count ≥ 0.5 x 109/L, Platelet count ≥ 100 x 109/L, Serum creatinine ≤ 2 mg/dL (0.18mmol/L), Serum bilirubin ≤ 2mg/dL (0.034mmol/L), Granulocyte count > 2.5x109/L, Aspartate Amino Transférase (ASAT), Alanine Amino Transferase (ALAT) < 2.5 x upper limit of normal, Activated Partial Thromboplastin Time (aPTT) within the normal ranges ±25%, Thromplastin (TP) ≥ 80%

Exclusion Criteria:

* Clinically significant heart disease.
* Serious illness, eg. serious infections requiring antibiotics, uncontrolled peptic ulcer, or central nervous system disorders.
* History of immunodeficiency disease or autoimmune disease.
* Metastatic disease to the central nervous system, unless treated and stable.
* Known HIV positivity.
* Known seropositivity for hepatitis B surface antigen.
* Concomitant treatment with steroids, antihistamine drugs. Topical or inhalation steroids are permitted.
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
* Pregnancy or lactation.
* Women of childbearing potential not using a medically acceptable means of contraception.
* Psychiatric or addictive disorders that may compromise the ability to give informed consent.
* Lack of availability of the patient for immunological and clinical follow-up assessment.
* Coagulation or bleeding disorders.
* Kidney dysfunction with creatinine > 2 X the upper limit of the normal value.
* Reported strong (allergic) reactions to previous vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Michielin, MD PhD, Principal Investigator — Oncology Department, Centre Hospitalier Universitaire Vaudois, Lausanne
Locations (1):
- Oncology Department, CHUV, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Sierro S, Romero P, Speiser DE. The CD4-like molecule LAG-3, biology and therapeutic applications. Expert Opin Ther Targets. 2011 Jan;15(1):91-101. doi: 10.1517/14712598.2011.540563. PMID 21142803
- [Background] Brignone C, Escudier B, Grygar C, Marcu M, Triebel F. A phase I pharmacokinetic and biological correlative study of IMP321, a novel MHC class II agonist, in patients with advanced renal cell carcinoma. Clin Cancer Res. 2009 Oct 1;15(19):6225-31. doi: 10.1158/1078-0432.CCR-09-0068. Epub 2009 Sep 15. PMID 19755389
- [Background] Speiser DE, Romero P. Molecularly defined vaccines for cancer immunotherapy, and protective T cell immunity. Semin Immunol. 2010 Jun;22(3):144-54. doi: 10.1016/j.smim.2010.03.004. Epub 2010 Apr 21. PMID 20413326
- [Result] Legat A, Maby-El Hajjami H, Baumgaertner P, Cagnon L, Abed Maillard S, Geldhof C, Iancu EM, Lebon L, Guillaume P, Dojcinovic D, Michielin O, Romano E, Berthod G, Rimoldi D, Triebel F, Luescher I, Rufer N, Speiser DE. Vaccination with LAG-3Ig (IMP321) and Peptides Induces Specific CD4 and CD8 T-Cell Responses in Metastatic Melanoma Patients--Report of a Phase I/IIa Clinical Trial. Clin Cancer Res. 2016 Mar 15;22(6):1330-40. doi: 10.1158/1078-0432.CCR-15-1212. Epub 2015 Oct 23. PMID 26500235
- See also: Multidisciplinary Oncology Center, CHUV, Lausanne — http://www.cancer-chuv.ch/ccl_home.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 patients were selected between June 15, 2010 and January 24, 2013. Among them 10 patients were included in the group 1 and 6 in the group 2. Since January 2013, 11 patients have been prescreened but could not be included in the study. On April 15, 2014, the decision had to taken to abort the study (16 patients included, while 28 were planned).
Pre-assignment Details: An unexplained high percentage, i.e. about 90% of the 11 prescreened patients were HLA-A2 negative. We assume that this was due to the increasing ethnic diversity of patients.
  The consequence of the time delay was that some of the peptides expired definitively.
Groups:
- Group 1: 2 vaccine injections in same limb (vaccine 1 : NY-ESO-1, MAGE-3.A2, NA-17 peptides + IMP321 + Montanide) (vaccine 2 : Melan-A, MAGE-A3-DP4 peptides + IMP321 + Montanide)
  2 vaccine injections in 1 limb: All participants receive the vaccine separated in 2 syringes with syringe 1 containing NA-17, MAGE-3.A2 and NY-ESO-1 peptides with IMP321/LAG3 ± Montanide, and syringe 2 containing Melan-A and MAGE-A3-DP4 peptides with IMP321/LAG-3 ± Montanide. The content of each syringe is injected s.c. in the same limb at about 5 cm distance from each other.
- Group 2: 2 vaccine injections in different limbs (vaccine 1: NY-ESO-1, MAGE-3.A2, NA-17 peptides + IMP321 + Montanide) (vaccine 2: Melan-A, MAGE-A3-DP4 peptides + IMP321 + Montanide)
  2 vaccine injections in different limbs: All participants receive the vaccine separated in 2 syringes with syringe 1 containing NA-17, MAGE-3.A2 and NY-ESO-1 peptides with IMP321/LAG3 ± Montanide, and syringe 2 containing Melan-A and MAGE-A3-DP4 peptides with IMP321/LAG-3 ± Montanide.The content of each syringe is injected s.c. in different limbs.
- Group 3: 2 vaccine injections in different limbs (vaccine 1: NY-ESO-1, MAGE-3.A2, NA-17 peptides + IMP321 + Montanide) (vaccine 2: Melan-A peptide + IMP321 + Montanide)
  2 vaccine injections in different limbs, the vaccine does not contain the MHC class II peptide MAGE-A3-DP4: All participants receive the vaccine separated in 2 syringes with syringe 1 containing NA-17, MAGE-3.A2 and NY-ESO-1 peptides with IMP321/LAG3 ± Montanide, and syringe 2 containing Melan-A peptide with IMP321/LAG-3 ± Montanide. The content of each syringe is injected s.c. in different limbs.
Period: Cycle 1
Arm/Group | Group 1 | Group 2 | Group 3
Started | 10 | 6 | 0
Completed | 10 | 6 | 0
Not Completed | 0 | 0 | 0
Period: Cycle 2
Arm/Group | Group 1 | Group 2 | Group 3
Started | 10 | 6 | 0
Completed | 10 | 5 | 0
Not Completed | 0 | 1 | 0
Period: Cycle 3
Arm/Group | Group 1 | Group 2 | Group 3
Started | 10 | 5 | 0
Completed | 10 | 4 | 0
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Due to premature trial termination, no patients could be enrolled in the Group 3.
Groups:
- Group 1: 2 Vaccine Injections in 1 Limb: 9 patients initially planned: patients received peptides with IMP321/LAG-3Ig and Montanide in 2 injections sites at 5 cm distance from each other 2 vaccine injections in same limb (vaccine 1 : NY-ESO-1, MAGE-3.A2, NA-17 peptides + IMP321 + Montanide)(vaccine 2 : Melan-A, MAGE-A3-DP4 peptides + IMP321 + Montanide)
  2 vaccine injections in 1 limb: Participants receive the vaccine separated in 2 syringes with syringe 1 containing NA-17, MAGE-3.A2 and NY-ESO-1 peptides with IMP321/LAG3 ± Montanide, and syringe 2 containing Melan-A and MAGE-A3-DP4 peptides with IMP321/LAG-3 ± Montanide. The content of each syringe is injected s.c. in the same limb at about 5 cm distance from each other.
- Group 2: 2 Injections in Different Limbs: 9 patients initially planned: patients received the same vaccine in 2 syringes injected each in a distinct limb 2 vaccine injections in different limbs (vaccine 1: NY-ESO-1, MAGE-3.A2, NA-17 peptides + IMP321 + Montanide) (vaccine 2: Melan-A, MAGE-A3-DP4 peptides + IMP321 + Montanide)
  2 vaccine injections in different limbs: Participants receive the vaccine separated in 2 syringes with syringe 1 containing NA-17, MAGE-3.A2 and NY-ESO-1 peptides with IMP321/LAG3 ± Montanide, and syringe 2 containing Melan-A and MAGE-A3-DP4 peptides with IMP321/LAG-3 ± Montanide.The content of each syringe is injected s.c. in different limbs.
- Group 3: 2 Injections in Different Limbs: 9 patients initially planned: due to premature trial termination, no patients could be enrolled in this last group. 2 vaccine injections in different limbs; patients of this group should have received the same vaccine but without the MHC class II peptide (MAGE-A3 LP) in 2 syringes injected each in a distinct limb.
  2 vaccine injections without MHC class II peptide in different limbs: Participants receive the vaccine separated in 2 syringes with syringe 1 containing NA-17, MAGE-3.A2 and NY-ESO-1 peptides with IMP321/LAG3 ± Montanide, and syringe 2 containing Melan-A peptide with IMP321/LAG-3 ± Montanide.
- Total: Total of all reporting groups
Arm/Group | Group 1: 2 Vaccine Injections in 1 Limb | Group 2: 2 Injections in Different Limbs | Group 3: 2 Injections in Different Limbs | Total
Number analyzed (Participants) | 10 | 6 | 0 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 0 | 10
  >=65 years | 5 | 1 | 0 | 6
Age, Continuous [Median (Full Range); unit: years] | 65.3 [53.5 to 84.4] | 50.2 [21.4 to 67.3] |  | 62.7 [21.4 to 84.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 |  | 8
  Male | 7 | 1 |  | 8
Region of Enrollment [Number; unit: participants]
  Switzerland | 10 | 6 |  | 16

OUTCOME MEASURES:

1. Primary Outcome: Ex Vivo Frequency of Melan-A Specific CD8+T Cells
Description: Cellular immunity was evaluated through the activation and the expansion of Melan-A-specific CD8+ cytotoxic T lymphocytes. Their frequency was measured in the peripheral blood mononuclear cells (PBMC) directly ex vivo (i.e. without prior in vitro expansion) by multicolor flow cytometry with Melan-A ELA tetramers.
  The fold change for each time point compared to baseline was calculated as: Melan-A-specific CD8+ T cell frequency at the time point/ Melan-A-specific CD8+ T cell frequency at baseline.
  Significant T cell response is defined by at least 2-fold change of Melan-A-specific CD8+ T cell frequency as compared to pre-immunotherapy.
Time Frame: Melan-A specific CD8+ T cells were measured in PBMC collected at the end of Cycle 1 (Week 7), end of Cycle 2 (Week 25), end of Cycle 3 (Week 40), and Follow-up (6 to 18 months after the end of Cycle 3).
Population: No patients were included in the group 3
Measure: Median (Standard Deviation); unit: Fold change of % Melan-A CD8+T ex vivo
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 10 | 6 | 0
Fold change of % Melan-A CD8+T ex vivo
  End cycle 1 | 1.21 (0.47) | 1.25 (1.44) |
  End cycle 2 | 1.09 (18.21) | 1.67 (2.14) |
  End cycle 3 | 0.91 (5.77) | 1.83 (1.79) |
  Follow up | 1.00 (2.14) | 0.28 (0.39) |
  Max | 1.21 (18.21) | 1.83 (2.14) |

2. Primary Outcome: In Vitro Frequency of MAGE A3.DP4-specific CD4+ T Cells Producing Interferon-gamma (IFN-γ)
Description: The activation of peptide-specific CD4+ T cells was analyzed in vitro before and after vaccination by Intracellular Cytokine Staining (ICS).
  From each patient, total CD4+ T-cells were stimulated in the presence of peptide MAGE-A3.DP4 LP (MAGE-A3243-258 peptide presented by autologous cells).
  After 10 days, cell cultures were challenged for 4h with the peptide or left unchallenged.
  Specific CD4+ T cells responses were identified via detection of IFN-γ producing cells.
Time Frame: MAGE A3.DP4 specific CD4+ T cells producing IFN-γ were measured in PBMC collected at the end of Cycle 1 (Week 7), end of Cycle 2 (Week 25), end of Cycle 3 (Week 40), and Follow-up (6 to 18 months after the end of Cycle 3).
Population: No patients were included in the group 3
Measure: Median (Standard Deviation); unit: % MAGE-A3.DP4 specific CD4+T IFN-γ
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 10 | 6 | 0
% MAGE-A3.DP4 specific CD4+T IFN-γ
  Baseline | 0 (0) | 0 (0) |
  End of cycle 1 | 0.47 (1.05) | 1.89 (2.23) |
  End of cycle 2 | 1.11 (1.06) | 1.63 (1.60) |
  End of cycle 3 | 2.00 (1.74) | 0.29 (0.91) |
  Follow up | 1.46 (1.97) | 0.77 (0.91) |

3. Primary Outcome: In Vitro Frequency of MAGE A3.DP4-specific CD4+ T Cells Producing Tumor Necrosis Factor-alpha (TNF-α)
Description: The activation of peptide-specific CD4+ T cells was analyzed in vitro before and after vaccination by ICS.
  From each patient, total CD4+ T-cells were stimulated in the presence of peptide MAGE-A3.DP4 LP (MAGE-A3243-258 peptide presented by autologous cells).
  After 10 days, cell cultures were challenged for 4h with the peptide or left unchallenged.
  Specific CD4+ T cells responses were identified via detection of TNF-α producing cells.
Time Frame: MAGE A3.DP4 specific CD4+ T-cells producing TNF-α were measured in PBMC collected at the end of Cycle 1 (Week 7), end of Cycle 2 (Week 25), end of Cycle 3 (Week 40), and Follow-up (6 to 18 months after the end of Cycle 3).
Population: No patients were included in the group 3
Measure: Mean (Standard Deviation); unit: % MAGE A3.DP4 specific CD4+T TNFα
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 10 | 6 | 0
% MAGE A3.DP4 specific CD4+T TNFα
  Baseline | 0.01 (0.01) | 0 (0) |
  End of cycle 1 | 0.70 (2.33) | 3.39 (2.35) |
  End of cycle 2 | 1.05 (2.74) | 2.31 (2.04) |
  End of cycle 3 | 1.63 (3.90) | 0.60 (0.80) |
  Follow up | 2.04 (1.57) | 3.63 (3.06) |

4. Primary Outcome: In Vitro Frequency of MAGE A3.DP4-specific CD4+ T Cells
Description: Frequencies of specific MAGE-A3.DP4-specific CD4+ T cells were quantified by flow cytometry using class II tetramers after 10 days of in vitro stimulation.
  The fold change for each time point compared to baseline was calculated as: MAGE-A3.DP4-specific CD4+ T cell frequency at the time point/ MAGE-A3.DP4-specific CD4+ T cell frequency at baseline.
Time Frame: MAGE A3.DP4 specific CD4+ T cells were measured in PBMC collected at the end of Cycle 1 (Week 7), end of Cycle 2 (Week 25), end of Cycle 3 (Week 40) and Follow-up (6 to 18 months after the end of Cycle 3).
Population: No patients were included in group 3
Measure: Median (Standard Deviation); unit: Fold change of % MageA3.DP4 CD4+T
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 10 | 6 | 0
Fold change of % MageA3.DP4 CD4+T
  End cycle 1 | 0.19 (2.02) | 0.22 (0.17) |
  End of cycle 2 | 0.88 (1.79) | 1.97 (1.77) |
  End of cycle 3 | 1.57 (1.64) | 0.66 (0.61) |
  Follow up | 0.63 (2.63) | 0.62 (0.32) |
  Max | 1.96 (2.67) | 1.28 (1.69) |

5. Primary Outcome: In Vitro Frequency of Melan-A-specific CD8+T Cells After Stimulation
Description: After 12 days of in vitro stimulation with Melan-A peptides, CD8+ T cells were analyzed by flow cytometry using tetramer staining.
  The fold change for each time point compared to baseline was calculated as: Melan-A-specific CD8+ T cell frequency at the time point/ Melan-A-specific CD8+ T cell frequency at baseline.
  Significant T cell response is defined by at least 2-fold change of Melan-A-specific CD8+ T cell frequency as compared to pre-immunotherapy.
Time Frame: In vitro stimulated Melan-A specific CD8+ T cells were measured in PBMC collected at the end of Cycle 1 (Week 7), end of Cycle 2 (Week 25), end of Cycle 3 (Week 40) and Follow-up (6 to 18 months after the end of Cycle 3).
Population: No patients were included in group 3
Measure: Median (Standard Deviation); unit: Fold change of % Melan-A CD8+T cells
Arm/Group | Group 1: 2 Vaccine Injections in 1 Limb | Group 2: 2 Injections in Different Limbs | Group 3: 2 Injections in Different Limbs
Number analyzed (Participants) | 10 | 6 | 0
Fold change of % Melan-A CD8+T cells
  End cycle 1 | 0.97 (3.75) | 2.60 (1.84) |
  End cycle 2 | 1.10 (4.61) | 5.33 (11.02) |
  End cycle 3 | 0.69 (9.57) | 2.84 (44.83) |
  Follow up | 2.83 (16.73) | 0 (0) |
  Max | 2.83 (16.73) | 5.33 (44.83) |

6. Primary Outcome: In Vitro Frequency of NY-ESO-1-specific CD8+ T Cells
Description: After 12 days of in vitro stimulation with NY-ESO-1 peptide, CD8+ T cells were analyzed by flow cytometry using tetramer staining.
  The fold change for each time point compared to baseline was calculated as: NY-ESO-1-specific CD8+ T cell frequency at the time point/ NY-ESO-1-specific CD8+ T cell frequency at baseline.
Time Frame: In vitro stimulated NY-EYO-1 specific CD8+ T cells were measured in PBMC collected at the end of Cycle 1 (Week 7), end of Cycle 2 (Week 25), end of Cycle 3 (Week 40), and Follow-up (6 to 18 months after the end of Cycle 3).
Population: No patients were included in the group 3
Measure: Median (Standard Deviation); unit: Fold change of % NY-ESO-1 CD8+T cells
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 10 | 6 | 0
Fold change of % NY-ESO-1 CD8+T cells
  End cycle 1 | 0.01 (0.45) | 0 (0) |
  End cycle 2 | 0 (0.3) | 0 (0.2) |
  End cycle 3 | 0.005 (0.23) | 0.06 (0.95) |
  Follow up | 0.02 (0.64) | 0 (0) |
  Max | 0.02 (0.64) | 0.06 (0.95) |

7. Secondary Outcome: Tumor Response
Description: The assessment of the baseline disease status was performed, using CT (Computed Tomography) scan or PET (Positron Emission Tomography)/ CT scan, at screening visit or within 8 weeks preceding the screening visit. Imagery examinations occurred after the end of each vaccination cycle. The tumor response was assessed according to the classification World Health Organization (WHO) 1979 and defined as:
  * No evidence of disease (NED),
  * Stable disease (SD): change in size of all measurable lesions (the sum of the products of the greatest and perpendicular parameters), of less than a 25% increase or 25% decrease from baseline for at least 4 weeks, without appearance of new lesions or progression of any lesion.
  * Progressive disease (PD): appearance of new tumors, or increase in size of any measurable tumor by at least 25% of the sum of the product of the greatest and perpendicular diameter.
Time Frame: Change from baseline in tumor response at the end of Cycle 1 (Week 7), end of Cycle 2 (Week 25) and end of Cycle 3 (Week 40)
Population: No patients were included in the group 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 10 | 6 | 0
Participants
  Disease status at cycle 1 end: NED | 7 | 5 |
  Disease status at cycle 1 end: SD | 0 | 0 |
  Disease status at cycle 1 end: PD | 3 | 1 |
  Disease status at cycle 2 end: number analyzed (Participants) | 10 | 5 | 0
  Disease status at cycle 2 end: NED | 8 | 4 |
  Disease status at cycle 2 end: SD | 0 | 0 |
  Disease status at cycle 2 end: PD | 2 | 1 |
  Disease status at cycle 3 end: number analyzed (Participants) | 10 | 4 | 0
  Disease status at cycle 3 end: NED | 8 | 4 |
  Disease status at cycle 3 end: SD | 0 | 0 |
  Disease status at cycle 3 end: PD | 2 | 0 |

ADVERSE EVENTS:
Time Frame: All adverse events were recorded from the first vaccination visit (Day 0) to the last vaccination visit (V9) of the cycle 3 of vaccination (week 39) therefore the adverse events were collected for 9 months.
Description: No patients were included in the group 3. All adverse events were collected irrespective of their frequency, their severity and relationship to the study drug.
  The adverse events that were expected, according to the Investigator's Brochure of the different vaccine components, were assessed systematically at each visit study.
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/6 | 0/0
Other Adverse Events (participants affected / at risk) | 10/10 | 6/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=10) | Group 2 (N=6) | Group 3 (N=0)
Upper limb fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=10) | Group 2 (N=6) | Group 3 (N=0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy inguinal (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 0 (0)
Lymphoedema (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0)
Haematoma (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 0 (0)
Diabetes mellitus (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eya lesions (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aphtous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (3) | 0 (0)
Asthenia (General disorders) | 4 (8) | 2 (6) | 0 (0)
Contusion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flush (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 2 (4) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (2) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (3) | 0 (0)
Performance status decreased (General disorders) | 1 (1) | 0 (0) | 0 (0)
Previous studies injection site induration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected lymphocele (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Increased lactade dehydrogenase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Karnofsky scale worsened (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocytes count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Positron emission abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urine leucocytes esterase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Abnormal weight gain (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extermity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Upper limb fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Malignat melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 1 (7) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Sinus polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizzines (Nervous system disorders) | 2 (2) | 1 (3) | 0 (0)
Headache (Nervous system disorders) | 5 (26) | 4 (8) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Cystitis/Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Balanitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Menauposal symptoms (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menstruation delayed (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis haemophilus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (6) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysponea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hoarsness of voice (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Capilaritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Erythema eyelid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Granuloma skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Puritus (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0 (0)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous nodules (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 10 (41) | 6 (42) | 0 (0)
Injection site induration (General disorders) | 10 (56) | 5 (44) | 0 (0)
Injection site pain (General disorders) | 10 (47) | 6 (25) | 0 (0)
Injection site recall reaction (General disorders) | 7 (15) | 3 (5) | 0 (0)
Injection site warmth (General disorders) | 4 (14) | 5 (24) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (12) | 1 (1) | 0 (0)
Asthenia (General disorders) | 4 (8) | 2 (6) | 0 (0)
Chills (General disorders) | 4 (16) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (26) | 4 (7) | 0 (0)
Influenza like illness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (4) | 1 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (15) | 1 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 1 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes